CLINICAL TRIAL: NCT05132478
Title: The Effect of Surgeon Emotional Support on Treatment Choice for Low-risk Thyroid Cancer: a Randomized Hypothetical Choice Experiment
Brief Title: The Effect of Surgeon Emotional Support on Treatment Choice for Low-risk Thyroid Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: UW21090; A539722 (Other: UW Madison); Protocol Version 11/8/2021 (Other: UW Madison); K08CA230204 (NIH); 2021-1079 (Other: UW Madison); NCI-2022-02184 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Results first posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Thyroid Cancer; Thyroid Nodule; Benign Thyroid Nodule
Keywords: thyroid cancer; low-risk; thyroidectomy; emotional support; treatment
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Video (Active Comparator): A video simulation of a patient-surgeon discussion about treatment options for low-risk thyroid cancer WITHOUT emotionally supportive statements
  Interventions: Other: Standard Video
- Emotionally Supportive Video (Experimental): A video simulation of a patient-surgeon discussion about treatment options for low-risk thyroid cancer WITH emotionally supportive statements
  Interventions: Other: Emotionally Supportive Video

INTERVENTIONS:
Other: Emotionally Supportive Video — The video is approximately 6 1/2 minutes in length and portrays an emotionally supportive conversation between a patient and surgeon during which the surgeon discusses: the diagnosis, prognosis, available treatment options, benefits and harms of the options, and need for decision making. The surgeon speaks for the majority of the simulated visit and discusses total and hemi-thyroidectomy with the addition of emotionally supportive statements and gestures.
  Arms: Emotionally Supportive Video
Other: Standard Video — The video is approximately 5 minutes in length and portrays a standard conversation between a patient and surgeon during which the surgeon discusses: the diagnosis, prognosis, available treatment options, benefits and harms of the options, and need for decision making. The surgeon speaks for the majority of the simulated visit and discusses total and hemi-thyroidectomy.
  Arms: Standard Video

SUMMARY:
118 adults with benign thyroid nodules who were seen at a UW Health clinic for a fine needle biopsy and do not need surgery will be enrolled and can expect to be on study for a one-time visit of up to 60 minutes. Each participant will be randomized to watch one of two videos simulating a patient-surgeon discussion about treatment options for low-risk thyroid cancer with or without emotionally supportive statements.

DETAILED DESCRIPTION:
In this study, the investigators will test the extent to which emotionally supportive communication from a surgeon is associated with patient preference for total thyroidectomy. The investigators will conduct a hypothetical choice experiment with "analogue" patients, defined as those with a benign thyroid nodule not requiring surgery.

Baseline measures will be collected, then participants will be randomized to watch a video simulation of a patient-surgeon discussion about treatment options for low-risk thyroid cancer with or without emotionally supportive statements.

The investigators hypothesize that increased emotionally supportive communication by the surgeon will decrease the likelihood of patients choosing total thyroidectomy, reduce anxiety and thyroid cancer fear, and increase decisional confidence, perceived physician empathy, trust in physician, and information recall.

ELIGIBILITY:
Inclusion Criteria (Determined during electronic medical record (EMR) screening):

* Seen in a UW Health Clinic for fine needle aspiration (FNA) of a thyroid nodule in the last 30 days
* Thyroid nodule measures ≤4 centimeters
* Benign thyroid nodule biopsy result
* Able to speak and read English
* Access to internet

Inclusion Criteria (Determined/reconfirmed during pre-study screening on Qualtrics):

* Seen in a UW Health Clinic for FNA of a thyroid nodule in the last 30 days

Exclusion Criteria (Determined during EMR screening):

* Additional thyroid nodule biopsy results that are not benign
* History of thyroid cancer
* History of thyroid surgery
* Has seen a surgeon about thyroid or parathyroid surgery
* Has a referral to see a surgeon about thyroid surgery
* Deaf
* Blind
* Vulnerable populations such as prisoners

Exclusion Criteria (Reconfirmed during pre-study screening on Qualtrics):

* History of thyroid cancer
* History of thyroid surgery
* Has seen a surgeon about thyroid or parathyroid surgery
* Plans to see a surgeon about thyroid surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corrine Voils, PhD, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected for this study will be transferred and analyzed at the University of Michigan. After the study is completed, the de-identified, archived data may be transmitted to and stored at a data repository for use by other researchers including those outside of the study. Permission to transmit data to the University of Michigan and data repository will be included in the informed consent.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the completion of the primary endpoint.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at the University of Wisconsin Carbone Cancer Center from November 2021 to February 2023
Pre-assignment Details: 555 patients were screened, 221 were deemed eligible and invited to participate, 128 consented, 2 participants discontinued after consent prior to randomization, 126 were randomized to start, 2 participants did not complete the survey, and 6 participants who completed the survey greater than 30 days past biopsy, were excluded because they did not meet the eligibility criteria of needing to be within 30 days of their biopsy.
Period: Overall Study
Arm/Group | Emotionally Supportive Video | Standard Video
Started | 64 | 62
Completed Survey | 63 | 61
Analysis Population (Excluded from analysis are those participants who completed the survey greater than 30 days past biopsy.) | 60 | 58
Completed | 60 | 58
Not Completed | 4 | 4
Not completed — did not complete survey after consent | 1 | 1
Not completed — excluded from analysis because survey was completed >30 days past biopsy | 3 | 3

BASELINE CHARACTERISTICS:
Population: Baseline information provided for analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Emotionally Supportive Video | Standard Video | Total
Number analyzed (Participants) | 60 | 58 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (14.3) | 56.7 (13.3) | 55.2 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 51 | 101
  Male | 10 | 7 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 55 | 56 | 111
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 54 | 50 | 104
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 60 | 58 | 118
Education Level [Count of Participants; unit: Participants]
  Some High School or Less | 0 | 1 | 1
  High School Graduate | 6 | 4 | 10
  Some College or Associate's Degree | 17 | 19 | 36
  Bachelor's Degree | 18 | 18 | 36
  Graduate or PhD | 19 | 14 | 33
  Unknown/Not Reported | 0 | 2 | 2
Number of Participants with Bilateral Nodules [Count of Participants; unit: Participants] | 29 | 25 | 54
Nodule Size [Count of Participants; unit: Participants] — Number of participants who self-reported that their largest nodule biopsied was in the size category indication: less than or equal to 2 cm, greater than 2 cm, or unknown (meaning that the patient did not know).
  Participants
    Less than or equal to 2 cm | 18 | 19 | 37
    Greater than 2 cm | 31 | 27 | 58
    Unknown | 11 | 12 | 23
Number of Participants with Symptomatic Nodule [Count of Participants; unit: Participants] — Participants were asked: Before your thyroid nodule(s) was biopsied, were you experiencing any symptoms from your thyroid nodule(s)? Symptoms might include problems with your swallowing, voice, or neck pressure.
  Participants | 12 | 10 | 22
Hypothyroidism [Count of Participants; unit: Participants] | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Treatment Choice
Description: The investigators will measure which treatment participants would choose if they were the patient with thyroid cancer in the video (total thyroidectomy or lobectomy) immediately after they finish watching the video.
Time Frame: post video intervention (up to 60 minutes during the only study visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Emotionally Supportive Video | Standard Video
Number analyzed (Participants) | 60 | 58
Participants
  Total Thyroidectomy | 54 | 51
  Lobectomy | 6 | 7
Statistical Analysis 1: Comparison: Emotionally Supportive Video vs Standard Video; Test type: Superiority; p = 0.720, Regression, Logistic

2. Secondary Outcome: Participant Decisional Confidence Score
Description: Decisional Confidence in treatment option is measured using a single-item 10-point Likert scale where 1 is 'not confident at all' and 10 is 'completely confident'
Time Frame: post video intervention (up to 60 minutes during the only study visit)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emotionally Supportive Video | Standard Video
Number analyzed (Participants) | 60 | 58
score on a scale | 7.6 (2.1) | 7.7 (1.9)
Statistical Analysis 1: Comparison: Emotionally Supportive Video vs Standard Video; Test type: Superiority; p = 0.743, t-test, 2 sided

3. Secondary Outcome: State Trait Anxiety Inventory Brief (STAI Brief) Score
Description: The STAI brief is a 6-item survey about how the participant is feeling in the moment (calm, tense, upset, relaxed, content, worried) scored on a 4 point likert scale. The total possible range of scores is 6 to 24 with higher scores indicating higher anxiety.
Time Frame: measured at baseline and after video intervention (during 1 day study visit)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emotionally Supportive Video | Standard Video
Number analyzed (Participants) | 60 | 58
score on a scale
  Baseline | 9.5 (3.6) | 8.8 (2.7)
  Post-Intervention | 12.1 (4.1) | 11.1 (3.9)
Statistical Analysis 1: Comparison: Emotionally Supportive Video vs Standard Video; baseline; Test type: Superiority; p = 0.228, t-test, 2 sided
Statistical Analysis 2: Comparison: Emotionally Supportive Video vs Standard Video; Post-Intervention; Test type: Superiority; p = 0.176, t-test, 2 sided

4. Secondary Outcome: Adapted Thyroid Cancer Fear Scale Score
Description: The adapted Thyroid Cancer Fear Scale is a 8-item survey originally designed to assess fear of breast cancer in patients undergoing cancer screening. Items are rated on a 5-point scale from strongly disagree (1) to strongly agree (5) with a total possible range of scores from 8-40 where higher scores indicate increased fear of cancer.
Time Frame: measured at baseline and after video intervention (during 1 day study visit)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emotionally Supportive Video | Standard Video
Number analyzed (Participants) | 60 | 58
score on a scale
  baseline | 26.0 (7.0) | 27.0 (5.5)
  Post-Intervention | 24.2 (7.4) | 25.4 (6.7)
Statistical Analysis 1: Comparison: Emotionally Supportive Video vs Standard Video; baseline; Test type: Superiority; p = 0.410, t-test, 2 sided
Statistical Analysis 2: Comparison: Emotionally Supportive Video vs Standard Video; Post-Intervention; Test type: Superiority; p = 0.351, ANOVA

5. Secondary Outcome: Adapted Jefferson Scale of Patient's Perceptions of Physician's Empathy Score
Description: This 5-question instrument assesses patient perceptions of physician empathy, scored on a 7-point Likert scale ranging from 'strongly disagree' (1) to 'strongly agree' (7). Items are summed, with a max score of 35, higher values indicate a perception of more empathy.
Time Frame: post video intervention (up to 60 minutes during the only study visit)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emotionally Supportive Video | Standard Video
Number analyzed (Participants) | 60 | 58
score on a scale | 34.5 (5.8) | 25.9 (9.1)
Statistical Analysis 1: Comparison: Emotionally Supportive Video vs Standard Video; Test type: Superiority; p < 0.001, t-test, 2 sided — calculated p-value

6. Secondary Outcome: Adapted Trust in Physician Scale Score
Description: This 5-question instrument assesses patient trust in a physician, scored on a 5-point Likert scale ranging from 'strongly disagree' (1) to 'strongly agree' (5). Responses are summed and scores are on a scale of 5 to 25, with higher values indicating more trust.
Time Frame: post video intervention (up to 60 minutes during the only study visit)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emotionally Supportive Video | Standard Video
Number analyzed (Participants) | 60 | 58
score on a scale | 12.0 (2.6) | 10.4 (3.1)
Statistical Analysis 1: Comparison: Emotionally Supportive Video vs Standard Video; Test type: Superiority; p < 0.001, t-test, 2 sided — calculated p-value

ADVERSE EVENTS:
Time Frame: This study involves one study visit that will take up to 60 minutes.
Description: The current study will pose minimal risk to the participants. Although no problems or adverse events are expected, any study related adverse events will be documented and reported to the local IRB per institutional policy.
Arm/Group | Emotionally Supportive Video | Standard Video
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/58
Other Adverse Events (participants affected / at risk) | 0/60 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT05132478/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT05132478/ICF_000.pdf